CLINICAL TRIAL: NCT05539716
Title: Metabolism and Sleep Apnea Treatment
Acronym: MaST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Naresh Punjabi, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20210670; 5R01HL146709-04 (NIH)
Record Dates: First submitted 2022-05-16; First posted 2022-09-14 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Obstructive Sleep Apnea; Fat Disorder
MeSH Terms: conditions — Sleep Apnea, Obstructive; Lipid Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- No Intervention (Aim 1) Group (No Intervention): Participants in this group will not receive an intervention and will only undergo several testing procedures conducted within 3 to 4 weeks to assess OSA severity.
- PAP Therapy and Lifestyle Intervention (Aim 2) Group (Experimental): Participants in the Aim 1 Group found to have moderate to severe OSA (defined as having a Apnea-Hypopnea Index (AHI) of 15.0 events/hour or more) randomized to this arm will receive the PAP therapy and Lifestyle Intervention for 12 weeks.
  Interventions: Device: PAP Therapy; Behavioral: Lifestyle Counseling Intervention
- Lifestyle Intervention Only (Aim 2) Group (Experimental): Participants in the Aim 1 Group found to have moderate to severe OSA (defined as having a Apnea-Hypopnea Index (AHI) of 15.0 events/hour or more) randomized to this arm will receive only the Lifestyle Intervention for 12 weeks.
  Interventions: Behavioral: Lifestyle Counseling Intervention

INTERVENTIONS:
Device: PAP Therapy — Auto-PAP device (ResMed AirsenseTM Autoset) with a heated humidifier will be provided along with an appropriate mask and connecting hose for nightly use
  Arms: PAP Therapy and Lifestyle Intervention (Aim 2) Group
Behavioral: Lifestyle Counseling Intervention — Lifestyle intervention will include counseling on (a) education on nutrition and exercise; and (b) behavioral support for identifying lifestyle change strategies and problem-solving barriers to improve the regularity and duration of sleep. This will be conducted using brochures on weight loss and sleep hygiene
  Arms: Lifestyle Intervention Only (Aim 2) Group; PAP Therapy and Lifestyle Intervention (Aim 2) Group

SUMMARY:
The purpose of this research study is to see if obstructive sleep apnea (OSA) is associated with abnormalities in fat metabolism. Through this research study, the Investigator will evaluate how fat is metabolized in people with and without sleep apnea, what substances the fat tissue releases, and how these substances might change the way the body uses energy and sugar.

ELIGIBILITY:
Aim 1 Group:

Inclusion criteria:

* Age between 18-70 years
* Ability to provide consent

Exclusion criteria

* Body Mass Index (BMI) > 40 kg/m2
* Prevalent myocardial infarction, coronary revascularization, heart failure, and stroke
* Type 1 or Type 2 diabetes mellitus
* Current or prior use of PAP or oral appliance therapy for OSA
* Use of oral corticosteroids
* Unstable medical conditions that may preclude enrollment in the protocol such as: uncontrolled angina and/or congestive heart failure, uncontrolled blood pressure or resistant hypertension, severe chronic obstructive pulmonary disease, cancer, and active psychiatric disease (e.g., major depression)
* Other sleep disorders (e.g., circadian rhythm disorder, self-reported habitual sleep duration < 6h)
* Use of supplemental oxygen during wakefulness or sleep
* Central sleep apnea, obesity hypoventilation syndrome or Cheyne-Stokes respiration based on the home sleep test
* Resting awake Oxygen Saturation (SpO2) < 90%

Aim 2 Group:

Inclusion criteria:

* Age between 18-70 years
* Ability to provide consent
* Moderate-to-severe OSA (AHI ≥ 15/h);
* Demonstration of Positive Airway Pressure (PAP) use of > 4 h/night on 70% of the nights during 1-week run-in period
* Successful completion of all of the procedures for Aim 1.

Exclusion criteria:

* BMI: ≥ 40 kg/m2
* Type 1 or Type 2 diabetes mellitus
* Current use of PAP or oral appliance therapy for OSA
* Commercial driver or report of motor vehicle accident or near-miss due to sleepiness within the 2 previous years
* Epworth sleepiness score of 18 or more
* Use of oral corticosteroids
* Participation in another clinical trial
* Unstable medical conditions that may preclude enrollment in the protocol such as: uncontrolled angina and/or congestive heart failure, uncontrolled blood pressure or resistant hypertension, severe chronic obstructive pulmonary disease, cancer, and active psychiatric disease (e.g., major depression)
* Other sleep disorders (e.g., circadian rhythm disorder, self-reported habitual sleep duration < 6h)
* Use of supplemental oxygen during wakefulness or sleep
* Central sleep apnea, obesity hypoventilation syndrome or Cheyne-Stokes respiration based on the home sleep test
* Resting awake SpO2 < 90%

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Whole body lipolysis rate | Up to 3 months
  Measured using the Intravenous Glucose Tolerance Test (IVGTT) in micromoles/L/min assessed at baseline and again at 3 months

SECONDARY OUTCOMES:
Free Fatty Acids (FFA) Oxidation Rate | Up to 3 months
  Measured using the IVGTT in micromoles/L/min assessed at baseline and again at 3 months
Adipocyte insulin resistance | Up to 3 months
  Measured using the IVGTT in micromoles-microunits/L-ml assessed at baseline and again at 3 months
Lipolysis suppression slope | Up to 3 months
  Measured using the IVGTT in micromoles/L-min assessed at baseline and again at 3 months
Free fatty acid rebound slope | Up to 3 months
  Measured using the IVGTT in micromoles/L-min assessed at baseline and again at 3 months
Free fatty acid insulin sensitivity parameter | Up to 3 months
  Measured using the IVGTT in (picomoles/L x min)^-1 assessed at baseline and again at 3 months
Insulin sensitivity | Up to 3 months
  Measured using the IVGTT in (milliunits/L x min)^-1 assessed at baseline and again at 3 months
Acute insulin response to glucose | Up to 3 months
  Measured using the IVGTT in (milliunits/L) x minute assessed at baseline and again at 3 months
Glucose effectiveness | Up to 3 months
  Measured using the IVGTT in per minute assessed at baseline and again at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Naresh Punjabi, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No